CLINICAL TRIAL: NCT02376257
Title: Improving Therapeutic Learning in Depression: Proof of Concept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Ph.D., Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21MH102646 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2015-03-03 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
Keywords: Cognitive behavior therapy (CBT); d-cycloserine (DCS); Modafinil
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 250 mg DCS (Active Comparator): Baseline assessment (week 1), two weekly sessions when 250mg DCS is administered, and final week (week 4) when retention is assessed.
  Interventions: Drug: 250 mg DCS
- 100 mg modafinil (Active Comparator): Baseline assessment (week 1), two weekly sessions when 100 mg modafinil is administered, and final week (week 4) when retention is assessed.
  Interventions: Drug: 100 mg Modafinil
- Placebo (Placebo Comparator): Baseline assessment (week 1), two weekly sessions when placebo is administered, and final week (week 4) when retention is assessed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 250 mg DCS — Drug
  Other Names: d-cycloserine
  Arms: 250 mg DCS
Drug: 100 mg Modafinil — Drug
  Arms: 100 mg modafinil
Drug: Placebo — Drug
  Arms: Placebo

SUMMARY:
Despite advances in both pharmacotherapy and psychotherapy for major depression, non-response and partial-response remain relatively common outcomes, motivating the search for new treatments. This study is concerned with the development of one such novel treatment, the augmentation of exposure-based cognitive-behavior therapy (CBT) with d-cycloserine (DCS).

DETAILED DESCRIPTION:
Investigators will study the efficacy of DCS for augmenting therapeutic learning relevant for the treatment of depression (i.e., outside the extinction learning where DCS has been shown to have success). Specifically, the study investigates the role of DCS in enhancing declarative memory in depressed individuals, as evaluated by standardized tests and the retention of cognitive therapy session material. Investigators will also study an active comparison agent, modafinil, which appears to offer cognitive enhancing effects among both sleep-deprived and non-sleep-deprived individuals, but also appears to have drug-state (e.g., mood and side) effects that are not characteristic of DCS augmentation. Therefore, drug-context effects may affect memory retention over time. Hence, the study will evaluate memory enhancement effects both during the period of drug action as well as one week later when no drug is taken. Overall, investigators will examine cognitive function and memory performance over 4 study sessions in 96 men and women with major depression, who, in a double-blind fashion, will be randomly assigned to either: (1) 250mg DCS, (2) 100mg modafinil, or (3) placebo administered on Study Weeks 2 and 3. The memory tests include both items unique to a given study week and memory tasks that are repeated over time that allow assessment of memory and retention effects across one-week periods.

ELIGIBILITY:
Inclusion Criteria:

* Must have a DSM diagnosis of major depression as determined by structured diagnostic interview
* Must be free of psychotropic medications other than serotonin selective reuptake inhibitors (SSRIs) for at least 2 weeks
* No current suicidal ideation
* Able to speak and understand English
* Must be between the ages of 18 and 65, inclusive
* Must be a male, or a female who is not of childbearing potential (i.e., surgically sterile, postmenopausal for at least 1 year) or who is non-pregnant, non-lactating and using a medically accepted method of contraception. Acceptable methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, hormonal contraceptives. A woman of childbearing potential who is not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the trial

Exclusion Criteria:

* A DSM diagnosis of dementia, neurodegenerative disease, or other organic mental disorder; substance use disorder other than nicotine or caffeine in the last 3 months; bulimia or anorexia within the last 3 months; lifetime history of psychotic disorder or, bipolar disorder, or developmental disorder;
* A diagnosis of organic brain syndrome, mental retardation, or other cognitive dysfunction that could interfere with a participants capacity to participate in CBT or to complete safety and efficacy assessments
* A history of seizures (apart from childhood febrile seizures) or head trauma causing ongoing cognitive impairment
* An uncontrolled, unstable clinically significant medical condition (e.g., renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic or cerebrovascular disease, or malignancy, or poorly controlled hypertension (> 150/90mmHg) that may interfere with the interpretation of safety and efficacy evaluations in the opinion of the study physician or investigator
* Medical illness including hypertension, cardiac disease, liver disease, pulmonary diseases, central nervous system disease, and epilepsy;
* Recent (1 year) suicidal attempts or current suicidal ideation
* For women, currently pregnant, plans to be pregnant in the next 2 months, or currently breastfeeding
* Treatment with phenytoin, isoniazid, or propranolol or known sensitivity to modafinil or cycloserine
* A history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment
* Use of psychotropic medication (including stimulants) other than SSRIs
* Current daily use of alcohol or regular binge alcohol use as determined on the medical screen
* Insufficient command of the English language (i.e., cannot carry on a conversation with an interviewer in the English language or read associated text)
* Receipt of CBT in the previous five years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Otto, Ph. D, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Otto MW, Lee J, Hofmann SG, Hearon BA, Smits JA, Rosenfield D, Fava M, Wright JH. Examining the efficacy of d-cycloserine to augment therapeutic learning in depression. Contemp Clin Trials. 2016 May;48:146-52. doi: 10.1016/j.cct.2016.03.009. Epub 2016 Apr 16. PMID 27094721

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 mg DCS: Randomized drug intervention was administered on two weekly sessions following baseline evaluation
  250 mg DCS: Drug
- 100 mg Modafinil: Randomized drug intervention was administered on two weekly sessions following baseline evaluation
  100 mg Modafinil: Drug
- Placebo: Randomized drug intervention was administered on two weekly sessions following baseline evaluation
  Placebo: Drug
Period: Overall Study
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Started | 13 | 12 | 11
Completed | 13 | 12 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 11 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 11 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (14.0) | 26.4 (8.1) | 27.7 (10.8) | 29.9 (11.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 5 | 5 | 4 | 14
  Female | 7 | 6 | 7 | 20
  Transgender | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 10 | 12 | 9 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 8 | 9 | 5 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Immediate Memory measured by the Hopkins Verbal Learning Task [Mean (Standard Deviation); unit: number of correctly recalled words] — The Hopkins Verbal Learning Test (HVLT) consists of a 12-item word list, composed of four words from each of the three semantic categories. The patient's free recall of the list is recorded. The same procedure is repeated for two more trials. The total recall score for the last trial was used as the baseline score and ranged from a minimum of zero to a maximum of 12 correct answers. Population: Data were obtained on 34 of the 36 participants.
  number of correctly recalled words
    number analyzed (Participants) | 12 | 12 | 10 | 34
    (all) | 8.5 (1.3) | 9.6 (1.1) | 9.6 (1.7) | 9.2 (1.4)
Digits backwards [Mean (Standard Deviation); unit: Number of correct trials] — The examiner reads a list of digits and asks that each digit be read backwards. After correct scores, longer lists of digits are then provided. The total number of correct trials is recorded with higher scores indicating better performance. Scores can range from 0 to 16. Population: Data were obtained for 33 of the 36 participants.
  Number of correct trials
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 8.3 (2.7) | 9.5 (2.5) | 11.3 (2.5) | 9.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Recall of Cognitive Therapy Content
Description: A modified Cognitive Therapy Awareness Scale (CTAS) was used to assess delayed memory for cognitive therapy content from the computerized CBT. Higher scores indicate better memory for CBT skills. Scores range from 0 to 40.
Time Frame: Week 2 and Week 3
Population: Data was missing for two participants.
Measure: Mean (Standard Deviation); unit: Number of correct units of information
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 12 | 12 | 10
Number of correct units of information
  Week 2 | 25.4 (2.9) | 26.8 (4.0) | 24.7 (4.0)
  Week 3 | 28.2 (4.2) | 29.7 (3.9) | 28.7 (5.4)

2. Primary Outcome: 1 Week Delayed Recall of Emotional Story Items
Description: 1 Week Delayed Recall of a Threat-Related Story. Scores can range from 0 to 74, with higher scores reflect greater memory for story items.
Time Frame: Week 2 and Week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 13 | 12 | 11
units on a scale
  Week 2 | 13.5 (10.4) | 21.3 (8.0) | 16.1 (9.5)
  Week 3 | 25.0 (13.9) | 37.3 (12.3) | 26.4 (11.9)

3. Primary Outcome: 1 Week Delayed Recall Logical Memory
Description: Higher scores reflect greater recall of Wechsler Memory Scale (WMS) Story B content assessed one week after last rehearsal. Possible scores range from 0 to 25.
Time Frame: Week 2 and Week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 13 | 12 | 11
units on a scale
  Week 2 | 1.8 (2.3) | 4.4 (4.3) | 5.0 (3.8)
  Week 3 | 9.5 (5.0) | 12.8 (5.5) | 13.6 (5.1)

4. Secondary Outcome: Logical Memory Immediate Recall
Description: Immediate Story Recall from the Wechsler Memory Scale Story B. Higher scores reflect greater recall of the story material from the previous week. Possible scores range from 0 to 25.
Time Frame: Week 1, Week 2, Week 3
Measure: Mean (Standard Deviation); unit: Number of story units recalled
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 13 | 12 | 11
Number of story units recalled
  Week 1 | 14.8 (4.3) | 17.1 (2.8) | 16.2 (4.7)
  Week 2 | 17.7 (3.4) | 17.8 (4.1) | 18.2 (2.9)
  Week 3 | 18.5 (3.0) | 21.5 (2.2) | 21.2 (2.9)

5. Secondary Outcome: Immediate Memory Measured by the Hopkins Verbal Learning Task
Description: The Hopkins Verbal Learning Test (HVLT) consists of a 12-item word list, composed of four words from each of the three semantic categories. The patient's free recall of the list is recorded. The same procedure is repeated for two more trials. The total recall score for the third trial was used as the recorded score and ranged from a minimum of zero to a maximum of 12 correct answers.
Time Frame: Baseline, Week 1, Week 2, Week 3
Population: Data is missing for two participants.
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 12 | 12 | 10
Number of words recalled
  Baseline | 8.5 (1.3) | 9.6 (1.1) | 9.6 (1.7)
  Week 1 | 7.8 (1.7) | 9.9 (1.2) | 9.4 (1.5)
  Week 2 | 8.7 (1.6) | 9.7 (1.3) | 9.6 (1.3)
  Week 3 | 8.8 (1.8) | 10.1 (1.1) | 9.4 (2.2)

6. Secondary Outcome: Immediate Recall of Emotional Story Items
Description: Immediate recall score of items from the Emotional Story presentation. Scores can range from 0 to 74, with higher scores reflect greater memory for story items.
Time Frame: Week 1, Week 2, Week 3
Measure: Mean (Standard Deviation); unit: Number of story units recalled
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 13 | 12 | 11
Number of story units recalled
  Week 1 | 22.4 (11.9) | 35.2 (9.4) | 32.2 (13.3)
  Week 2 | 34.4 (12.6) | 46.8 (10.9) | 35.5 (11.0)
  Week 3 | 38.4 (12.9) | 49.9 (12.4) | 43.4 (11.3)

7. Secondary Outcome: Skills of Cognitive Therapy
Description: This measure assesses the self-reported use of skills from cognitive therapy. Scores can range from 8 to 40, and higher scores indicate greater use.
Time Frame: Week 2 and Week 3
Population: Data is missing for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 11 | 12 | 10
units on a scale
  Week 2 | 23.3 (6.4) | 20.5 (5.5) | 24.8 (5.6)
  Week 3 | 26.4 (8.5) | 24.3 (7.2) | 25.7 (4.4)

8. Secondary Outcome: Digits Backward
Description: The examiner reads a list of digits and asks that each digit be read backwards. The score is the total number of trials completed correctly; scores range from 0 to 16. Higher scores indicate better performance.
Time Frame: Baseline, Week 1, Week 2, Week 3
Population: Data is missing for two participants.
Measure: Mean (Standard Deviation); unit: Number of correct trials
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
Number analyzed (Participants) | 12 | 11 | 10
Number of correct trials
  Baseline | 8.3 (2.7) | 9.5 (2.5) | 11.3 (2.5)
  Week 1 | 9.25 (2.8) | 10.4 (2.2) | 12.2 (2.2)
  Week 2 | 10.0 (3.2) | 11.3 (2.0) | 12.1 (1.7)
  Week 3 | 9.6 (2.7) | 11.4 (2.2) | 11.7 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events for the visits on which study drugs were administered were assessed at the end of that session and (retrospectively) one week later for events occurring within several hours after that session (at Weeks 2 and 3, and retrospectively at 4). Serious adverse events were reported for the 4-week trial period as a whole.
Description: Adverse events were assessed by open query
Arm/Group | 250 mg DCS | 100 mg Modafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 4/13 | 7/12 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg DCS (N=13) | 100 mg Modafinil (N=12) | Placebo (N=11)
Increased Energy/Concentration (General disorders) | 2 (3) | 4 (5) | 2 (3) — Mild levels of symptoms reported with no distress
Fatigue/Low Motivation (General disorders) | 2 (3) | 3 (3) | 5 (5) — Mild levels of symptoms were reported with no distress

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-11-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02376257/Prot_000.pdf
  • Statistical Analysis Plan (2013-11-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02376257/SAP_001.pdf